CLINICAL TRIAL: NCT00803205
Title: A Phase 3 Efficacy and Safety Study of PTC124 as an Oral Treatment for Nonsense-Mutation-Mediated Cystic Fibrosis
Brief Title: Study of Ataluren (PTC124™) in Cystic Fibrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PTC124-GD-009-CF; Orphan Product Grant #FD003715 (Other Grant/Funding Number: Funding Source - FDA OOPD); 2008-003924-52 (EudraCT Number)
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Results first posted 2020-05-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; Nonsense mutation; Premature stop codon; PTC124; Ataluren; PTC Therapeutics
MeSH Terms: conditions — Cystic Fibrosis | interventions — ataluren

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ataluren (Experimental): Participants will receive ataluren 3 times per day (TID): 10 milligrams (mg)/kilogram (kg) of body weight with breakfast, 10 mg/kg with lunch, and 20 mg/kg with dinner (total daily dose 40 mg/kg). Treatment will continue for 48 weeks, after which participants will be followed for 4 weeks.
  Interventions: Drug: Ataluren
- Placebo (Placebo Comparator): Participants will receive placebo TID: 10 mg/kg of body weight with breakfast, 10 mg/kg with lunch, and 20 mg/kg with dinner (total daily dose 40 mg/kg). Treatment will continue for 48 weeks, after which participants will be followed for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ataluren — Ataluren will be provided as a vanilla-flavored powder to be mixed with water.
  Other Names: PTC124
  Arms: Ataluren
Drug: Placebo — Placebo matching to ataluren will be provided.
  Arms: Placebo

SUMMARY:
Cystic fibrosis (CF) is a genetic disorder caused by a mutation in the gene that makes the cystic fibrosis transmembrane conductance regulator (CFTR) protein. A specific type of mutation called a nonsense (premature stop codon) mutation is the cause of CF in approximately 10% of patients with the disease. Ataluren is an orally delivered investigational drug that has the potential to overcome the effects of the nonsense mutation. This study is a Phase 3 trial that will evaluate the clinical benefit of ataluren in adult and pediatric participants with CF due to a nonsense mutation. The main goals of the study are to understand whether ataluren can improve pulmonary function and whether the drug can safely be given for a long period of time. The study will also assess the effects of ataluren on CF pulmonary exacerbation frequency, cough frequency, health-related quality of life, antibiotic use for CF-related infections, CF-related disruptions to daily living, body weight, and CF pathophysiology.

DETAILED DESCRIPTION:
This study is a Phase 3, multicenter, randomized, double-blind, placebo-controlled, efficacy and safety study, designed to document the clinical benefit of ataluren when administered as therapy of participants with CF due to a nonsense mutation (premature stop codon) in the CFTR gene. It is planned that ~208 participants who are ≥6 years of age and have a forced expiratory volume in 1 second (FEV1) ≥40% and ≤90% of predicted will be enrolled. Study participants will be enrolled at sites in North America, Europe, and Israel. They will be randomized in a 1:1 ratio to either ataluren or placebo. Participants will receive study drug 3 times per day (at morning, midday, and evening) for 48 weeks. Participants will be evaluated at clinic visits every 8 weeks. Additional safety laboratory testing, which may be performed at the investigational site or at an accredited local laboratory or clinic, is required every 4 weeks for the first 6 months of study participation. At the completion of blinded treatment, all compliant participants will be eligible to receive open-label ataluren in a separate extension study.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent (parental/guardian consent and participant assent if <18 years of age)
* Age ≥6 years
* Body weight ≥16 kg
* Abnormal nasal transepithelial potential difference (TEPD) total chloride conductance (a less electrically negative value than -5 millivolts (mV) for total chloride conductance [Δchloride-free+isoproterenol])
* Sweat chloride >40 milliequivalents/liter (mEq/L)
* Documentation of the simultaneous presence of a nonsense mutation in at least 1 allele of the CFTR gene and a CF-causing mutation in the other CFTR allele, as determined by gene sequencing from a laboratory certified by the College of American Pathologists (CAP), under the Clinical Laboratory Improvement Act/Amendment (CLIA), or by an equivalent organization
* Verification that a blood sample has been drawn for confirmation of the presence of a nonsense mutation in the CFTR gene
* Ability to perform a valid, reproducible spirometry test using the study-specific spirometer with demonstration of an FEV1 ≥40% and ≤90% of predicted for age, gender, and height
* Resting oxygen saturation (as measured by pulse oximetry) ≥92% on room air
* Documentation by VivoMetrics that the participant has satisfactorily completed a 24-hour LifeShirt® cough frequency assessment
* Confirmed screening laboratory values within the central laboratory ranges (hepatic, adrenal, renal, serum electrolytes, and reproduction [women only] parameters)
* In participants who are sexually active, willingness to abstain from sexual intercourse or employ a barrier or medical method of contraception during the study drug administration and 4-week follow-up period
* Willingness and ability to comply with scheduled visits, drug administration plan, study restrictions, and study procedures

Exclusion Criteria:

* Known hypersensitivity to any of the ingredients or excipients of the study drug
* Any change (initiation, change in type of drug, dose modification, schedule modification, interruption, discontinuation, or reinitiation) in a chronic treatment/prophylaxis regimen for CF or for CF-related conditions within 4 weeks prior to start of study treatment
* Exposure to another investigational drug within 4 weeks prior to start of study treatment
* Treatment with systemic aminoglycoside antibiotics at the time of the Baseline TEPD assessment
* Treatment with intravenous antibiotics within 3 weeks prior to start of study treatment
* History of solid organ or hematological transplantation
* Ongoing immunosuppressive therapy (other than corticosteroids)
* Ongoing warfarin, phenytoin, or tolbutamide therapy
* Ongoing participation in any other therapeutic clinical trial
* Major complications of lung disease (including massive hemoptysis, pneumothorax, or pleural effusion) within 8 weeks prior to start of study treatment
* Evidence of pulmonary exacerbation or acute upper or lower respiratory tract infection (including viral illnesses) within 3 weeks prior to randomization
* Known portal hypertension
* Positive hepatitis B surface antigen, hepatitis C antibody test, or human immunodeficiency virus (HIV) test
* Pregnancy or breast-feeding
* Current smoker or a smoking history of ≥10 pack-years (number of cigarette packs/day * number of years smoked)
* Prior or ongoing medical condition (for example, concomitant illness, alcoholism, drug abuse, psychiatric condition), medical history, physical findings, electrocardiography findings, or laboratory abnormality that, in the Investigator's opinion, could adversely affect the safety of the participant, makes it unlikely that the course of treatment or follow-up would be completed, or could impair the assessment of study results.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2009-09-08 (Actual); Primary Completion 2011-11-12 (Actual); Study Completion 2011-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Temitayo Ajayi, MD, Study Director — PTC Therapeutics
Locations (38):
- United States (21):
  - University of Alabama-Birmingham, Birmingham, Alabama
  - Miller Children's Hospital Long Beach, Long Beach, California
  - Lucile Packard Children's Hospital, Palo Alto, California
  - Stanford, Palo Alto, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - The Children's Hospital, Aurora, Colorado
  - University of Miami, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Emory University Cystic Fibrosis Center, Atlanta, Georgia
  - Children's Memorial Hospital, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins Children's Center, Baltimore, Maryland
  - Children's Hospital Boston, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Beth Israel Medical Center, New York, New York
  - New York Medical College, Valhalla, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Rainbow Babies & Children's Hospital, Cleveland, Ohio
  - Childrens Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas, Tyler, Texas
  - University of Washington, Seattle, Washington
- Belgium (4):
  - Hôpital Erasme, Brussels
  - Hôpital Universitaire des Enfants Reine Fabiola, Brussels
  - University Hospital Brussels, Brussels
  - University Hospital Leuven, Leuven
- University of Toronto, Toronto, Canada
- France (3):
  - Hôpital Cochin, Paris
  - Hôpital Necker - Enfants Malades, Paris
  - Hôpital des Enfants, Toulouse
- Klinikum der Universität Köln, Cologne, Germany
- Hadassah University Hospital - Mount Scopus, Jerusalem, Israel
- Italy (2):
  - Università La Sapienza, Rome
  - Azienda Ospedaliera di Verona, Verona
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands
- Hospital Universitario La Paz, Madrid, Spain
- Karolinska University Hospital, Huddinge, Stockholm, Sweden
- United Kingdom (2):
  - Belfast City Hospital, Belfast
  - Alder Hey Children's Hospital, Liverpool

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kerem E, Konstan MW, De Boeck K, Accurso FJ, Sermet-Gaudelus I, Wilschanski M, Elborn JS, Melotti P, Bronsveld I, Fajac I, Malfroot A, Rosenbluth DB, Walker PA, McColley SA, Knoop C, Quattrucci S, Rietschel E, Zeitlin PL, Barth J, Elfring GL, Welch EM, Branstrom A, Spiegel RJ, Peltz SW, Ajayi T, Rowe SM; Cystic Fibrosis Ataluren Study Group. Ataluren for the treatment of nonsense-mutation cystic fibrosis: a randomised, double-blind, placebo-controlled phase 3 trial. Lancet Respir Med. 2014 Jul;2(7):539-47. doi: 10.1016/S2213-2600(14)70100-6. Epub 2014 May 15. PMID 24836205
- [Derived] Aslam AA, Sinha IP, Southern KW. Ataluren and similar compounds (specific therapies for premature termination codon class I mutations) for cystic fibrosis. Cochrane Database Syst Rev. 2023 Mar 3;3(3):CD012040. doi: 10.1002/14651858.CD012040.pub3. PMID 36866921

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 299 male and female participants with nonsense-mutation-mediated cystic fibrosis (nmCF) aged ≥6 years signed the informed consent form and were screened for eligibility, of which 61 did not meet entry criteria to participate in the study.
Pre-assignment Details: A total of 238 participants were randomized in a 1:1 ratio to either ataluren or placebo. Six participants (4 in the ataluren arm; 2 in the placebo arm) were excluded from the Intent-to-Treat (ITT) population because they did not have at least 1 post-Baseline forced expiratory volume (FEV1) assessment by Week 8.
Groups:
- Ataluren: Participants received ataluren 3 times daily (TID): 10 milligrams/kilogram (mg/kg) of body weight with breakfast, 10 mg/kg with lunch, and 20 mg/kg with dinner (total daily dose 40 mg/kg). Treatment continued for 48 weeks, after which participants were followed for 4 weeks.
- Placebo: Participants received placebo TID: 10 mg/kg of body weight with breakfast, 10 mg/kg with lunch, and 20 mg/kg with dinner (total daily dose 40 mg/kg). Treatment continued for 48 weeks, after which participants were followed for 4 weeks.
Period: Overall Study
Arm/Group | Ataluren | Placebo
Started | 120 | 118
Completed Week 16 | 107 | 113
Completed Week 24 | 103 | 110
As-Treated Population* (Randomized participants who received at least 1 dose of study drug *assessed for safety) | 120 | 118
ITT Population (Randomized participants with FEV1 data at Baseline and 1 post-Baseline assessment by Week 8) | 116 | 116
Per Protocol Population (Randomized participants who completed study treatment and had FEV1 data at Week 48) | 100 | 103
Completed | 100 | 104
Not Completed | 20 | 14
Not completed — Adverse Event | 7 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 9 | 9
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Medical Monitor Decision | 1 | 0
Not completed — Acquired a Lung Infection | 0 | 1
Not completed — Sponsor Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: The As-Treated Population: all randomized participants who received at least 1 dose of study drug.
Groups:
- Ataluren: Participants received ataluren TID: 10 mg/kg of body weight with breakfast, 10 mg/kg with lunch, and 20 mg/kg with dinner (total daily dose 40 mg/kg). Treatment continued for 48 weeks, after which participants were followed for 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Ataluren | Placebo | Total
Number analyzed (Participants) | 120 | 118 | 238
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.0 (10.06) | 23.2 (9.24) | 23.1 (9.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 59 | 117
  Male | 62 | 59 | 121

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Predicted Function (Percent-Predicted) of Forced Expiratory Volume in One Second (FEV1) at Baseline
Description: Spirometry was used to assess pulmonary function by measuring the percentage of predicted function, which was determined on the basis of the height value obtained at the same study visit, for FEV1 (the amount of air that can be exhaled in 1 second). Spirometry was assessed by using current guidelines of the American Thoracic Society (ATS) and European Respiratory Society (ERS). Baseline was the average of percent-predicted FEV1 at screening and randomization.
Time Frame: Baseline (Week 1)
Population: The ITT Population: all randomized participants with data for FEV1 at Baseline and a minimum of 1 post-Baseline assessment before Week 8. Here, 'Number analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of predicted FEV1
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 116 | 116
percentage of predicted FEV1 | 62.092 (13.6159) | 60.232 (15.1437)
Statistical Analysis 1: Comparison: Ataluren vs Placebo; Test type: Superiority; p = 0.3264, ANOVA

2. Primary Outcome: Percentage Change From Baseline in Percent-Predicted of FEV1 at Week 48
Description: Spirometry was used to assess pulmonary function by measuring the percentage of predicted function, which was determined on the basis of the height value obtained at the same study visit, for FEV1 (the amount of air that can be exhaled in 1 second). Spirometry was assessed by using current guidelines of the American Thoracic Society (ATS) and European Respiratory Society (ERS). The percentage of change in percent-predicted of FEV1 was calculated as follows: ([percent-predicted FEV1-Baseline percent-predicted FEV1]/Baseline percent-predicted FEV1)*100. Baseline was the average of percent-predicted FEV1 at screening and randomization. A negative change from Baseline indicates that percent-predicted of FEV1 decreased.
Time Frame: End of Treatment (EOT) (Week 48)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 116 | 116
percent change | -2.534 (13.2452) | -5.500 (12.5595)
Statistical Analysis 1: Comparison: Ataluren vs Placebo; Least squares (LS) mean estimates based on mixed model for repeated measures (Weeks 8, 16, 24, 32, 40 and 48) of relative change in percent-predicted FEV1 as the dependent variable; independent variables including Baseline percent-predicted FEV1, treatment, visit, interactions between treatment and visit and between Baseline percent-predicted FEV1 and visit; and stratification factors of Baseline age, Baseline inhaled antibiotics, and Baseline percent-predicted FEV1; Test type: Superiority; p = 0.1235, Mixed Models Analysis — The p-value is the LS-mean for the comparison between active treatment and placebo. The level of significance was 0.04998; Mean Difference (Final Values) = 2.7540, 95% CI 2-sided [-0.7560 to 6.2640], Standard Error of Mean 1.78124

3. Secondary Outcome: Rate of Pulmonary Exacerbations as Defined by Modified Fuch's Criteria Over 48 Weeks
Description: A Respiratory Event Form, which collected data on various signs, symptoms, and effects for each event, was completed by the Investigator when informed by the participant of a respiratory event. Pulmonary exacerbations were assessed by using the modified Fuchs' criteria, which defines an exacerbation as a respiratory event requiring treatment with parenteral antibiotics for any 4 of the following 12 symptoms, with or without intravenous antibiotics: change in sputum; new or increased hemoptysis; increased cough; increased dyspnea; fatigue; temperature >38°C; anorexia; sinus pain; change in sinus discharge; change in physical examination of the chest; decrease in pulmonary function by 10% or more from a previously recorded value; or radiographic changes indicative of pulmonary function. The 48-week exacerbation rate was determined by adding the weekly rates for each arm and dividing the sum by 48.
Time Frame: Baseline to EOT (Week 48)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: exacerbations
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 116 | 116
exacerbations | 1.42 [1.05 to 1.79] | 1.78 [1.38 to 2.17]

4. Secondary Outcome: Change From Baseline in Awake Cough Hourly Rate at Week 48
Description: The frequency of awake cough was measured using the LifeShirt, which incorporates motion-sensing transducers, electrodes, a microphone, and a 3-axis accelerometer into a lightweight vest. The rate was determined by dividing the total number of coughs by 24 (the number of hours of the observation period). Baseline was the latest, valid assessment prior to the treatment. A negative change from Baseline indicates that coughing decreased.
Time Frame: Baseline, EOT (Week 48)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: coughs/hour
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 116 | 116
coughs/hour
  Baseline: number analyzed (Participants) | 115 | 114
  Baseline | 28.218 (20.2726) | 24.472 (16.7828)
  Change From Baseline: number analyzed (Participants) | 97 | 100
  Change From Baseline | -0.595 (18.3221) | 0.882 (14.3936)

5. Secondary Outcome: Change From Baseline in the Respiratory Domain Score of the Revised Cystic Fibrosis Questionnaire (CFQ-R) at Week 48
Description: The CFQ-R consists of 44 items, including generic scales of physical functioning, role functioning, vitality, health perceptions, emotional functioning, and social functioning, and CF-specific scales of respiratory and digestive symptoms, body image, eating disturbances, and treatment burden. Each domain score ranges from 1 to 4. Scores were linearly transformed to a 0 to 100 scale, with higher scores indicating better health. Domain scores were calculated by using the following formula: 100 * (sum of responses - minimum possible sum)/ (maximum possible sum - minimum possible sum). The minimum possible sum = number of questions * 1; the maximum possible = the number of questions * 4. Baseline was the latest, valid assessment prior to the treatment. A negative change from Baseline indicates that health has worsened. Participants may have switched age groups during the study.
Time Frame: Baseline, EOT (Week 48)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 116 | 116
units on a scale
  Aged 6-13 years, Baseline: number analyzed (Participants) | 18 | 13
  Aged 6-13 years, Baseline | 77.78 (11.070) | 79.49 (16.879)
  Aged 6-13 years, Change From Baseline: number analyzed (Participants) | 12 | 7
  Aged 6-13 years, Change From Baseline | -0.69 (12.028) | -3.57 (21.973)
  Age ≥14 years , Baseline: number analyzed (Participants) | 95 | 101
  Age ≥14 years , Baseline | 70.06 (15.678) | 65.95 (16.771)
  Age ≥14 years, Change From Baseline: number analyzed (Participants) | 81 | 92
  Age ≥14 years, Change From Baseline | -2.81 (18.365) | -3.32 (16.245)

6. Secondary Outcome: Percent-Predicted of Forced Vital Capacity (FVC) at Baseline
Description: Spirometry was used to assess pulmonary function by measuring the percentage of predicted function, which was determined on the basis of the height value obtained at the same study visit, for FVC (the amount of air that can be exhaled after taking a deep breath). Spirometry was assessed by using current guidelines of the ATS and ERS. Baseline was the average of percent-predicted FVC at screening and randomization.
Time Frame: Baseline (Week 1)
Population: The ITT Population: all randomized participants with data for FEV1 at Baseline and a minimum of 1 post-Baseline assessment before Week 8. Here, 'Number analyzed 'signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of predicted FVC
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 116 | 116
percentage of predicted FVC | 78.332 (13.1825) | 76.609 (13.3711)

7. Secondary Outcome: Percentage Change From Baseline in Percent-Predicted of FVC at Week 48
Description: Spirometry was used to assess pulmonary function by measuring the percentage of predicted function, which was determined on the basis of the height value obtained at the same study visit, for FVC (the amount of air that can be exhaled after taking a deep breath). Spirometry was assessed by using current guidelines of the ATS and ERS. The percentage of change in percent-predicted of FVC was calculated as follows: ((percent-predicted FVC-Baseline percent-predicted FVC)/Baseline percent-predicted FVC)*100. Baseline was the average of percent-predicted FVC at screening and randomization. A negative change from Baseline indicates that percent-predicted of FVC decreased.
Time Frame: EOT (Week 48)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 116 | 116
percent change | -2.139 (10.0463) | -3.484 (9.9304)

8. Other Pre Specified Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAE)
Description: A TEAE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship that occurred or worsened in the period extending from first dose of study drug to 4 weeks after the last dose of study drug. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both SAEs and non-serious AEs. AE severity was graded as follows: Grade 1: mild; Grade 2: moderate; Grade 3: severe; Grade 4: life-threatening; Grade 5: fatal. A TEAE was considered related if in the opinion of the Investigator it was possibly or probably caused by the study drug. A summary of other non-serious AEs and all SAEs, regardless of causality is located in the Adverse Events module.
Time Frame: Baseline up to 4 Weeks Post-Treatment (Week 52) or Premature Discontinuation (PD)
Population: The As-Treated Population: all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percent of participants
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 120 | 118
percent of participants
  At least 1 TEAE | 98.3 | 97.5
  Grade 1 TEAE | 15.0 | 16.9
  Grade 2 TEAE | 67.5 | 55.1
  Grade 3 TEAE | 15.8 | 25.4
  Grade 4 TEAE | 0 | 0
  Grade 5 TEAE | 0 | 0
  Unrelated TEAE | 25.0 | 35.6
  Unlikely related TEAE | 32.5 | 26.3
  Possibly related TEAE | 28.3 | 29.7
  Probably related TEAE | 12.5 | 5.9
  Discontinuation due to TEAE | 6.7 | 2.5
  Serious TEAE | 37.5 | 40.7

9. Other Pre Specified Outcome: Rate of Study Drug Compliance by Drug Accountability
Description: Study drug compliance was assessed by using a Pharmacy Subject Study Drug Accountability Log (completed by the investigational site personnel). The rate of compliance was defined as 100 * (number of sachets taken/number of planned sachets) during the study. All calculations were based on the records of the first dose date to the last dose date. To differentiate dose strengths while maintaining the blind, each kit had a unique kit number and had prominent lettering "A" and "B." Each kit contained 65 packets of 1 of the dose strengths (125, 250, or 1000 mg or matching placebo). Labeling for active drug and placebo was identical.
Time Frame: Baseline up to EOT (Week 48)
Population: The As-Treated Population: all randomized participants who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: percent of doses taken
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 120 | 118
percent of doses taken
  Drug Kit A | 90.149 [18.24 to 109.24] | 85.119 [28.36 to 125.79]
  Drug Kit B | 90.830 [13.27 to 116.67] | 86.614 [25.22 to 107.60]

10. Other Pre Specified Outcome: Rate of Study Drug Compliance by Patient-Reported Data
Description: Patient-reported data were obtained from the participant's electronic daily diary, which was completed by the participant or the caregiver. During study treatment, the electronic daily diary was to be completed by the participant or caregiver each day for each dose. For each participant, compliance is described in terms of the percentage of study drug actually taken. All calculations were based on the records of the first dose date to the last dose date. To differentiate dose strengths while maintaining the blind, each kit had a unique kit number and had prominent lettering "A" and "B." Each kit contained 65 packets of 1 of the dose strengths (125, 250, or 1000 mg or matching placebo). Labeling for active drug and placebo was identical.
Time Frame: Baseline up to EOT (Week 48)
Population: The As-Treated Population: all randomized participants who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: percent of doses taken
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 120 | 118
percent of doses taken | 71.48 [0 to 98.5] | 69.27 [6.4 to 98.9]

11. Other Pre Specified Outcome: Concentration of Ataluren
Description: Blood samples were drawn immediately before administration of the first daily dose (dose taken with breakfast) of study drug and 2 hours after the first daily dose. Whenever possible, the pre-dose sample was to be obtained within 15 minutes of drug administration. Participants in the Placebo arm did not receive Ataluren and are not included in this Outcome Measure.
Time Frame: Predose and 2 Hours Postdose at Week 1, Week 16, Week 32, EOT (Week 48)
Population: The As-Treated Population: all randomized participants who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: micrograms/milliliter (ug/mL)
Arm/Group | Ataluren
Number analyzed (Participants) | 120
micrograms/milliliter (ug/mL)
  Week 1 Predose: number analyzed (Participants) | 119
  Week 1 Predose | 0 [0 to 0]
  Week 1 Postdose: number analyzed (Participants) | 117
  Week 1 Postdose | 14.100 [1.42 to 56.40]
  Week 16 Predose: number analyzed (Participants) | 103
  Week 16 Predose | 4.350 [0 to 52.60]
  Week 16 Postdose: number analyzed (Participants) | 104
  Week 16 Postdose | 11.900 [0.80 to 41.90]
  Week 32 Predose: number analyzed (Participants) | 99
  Week 32 Predose | 4.630 [0 to 29.20]
  Week 32 Postdose: number analyzed (Participants) | 97
  Week 32 Postdose | 13.400 [2.37 to 36.30]
  Week 48 Predose: number analyzed (Participants) | 97
  Week 48 Predose | 3.970 [0 to 27.00]
  Week 48 Postdose: number analyzed (Participants) | 96
  Week 48 Postdose | 10.500 [0 to 39.10]

12. Other Pre Specified Outcome: Rate of Interventions for Respiratory Symptoms
Description: During treatment, any intervention including hospitalization or use of oral, inhaled, or intravenous antibiotics was documented if it was due to an exacerbation-like episode. Participants and caregivers recorded interventions in an electronic diary. The rate of interventions was defined as the total days with interventions divided by the total study duration.
Time Frame: Baseline up to EOT (Week 48)
Population: The ITT Population: all randomized participants with data for FEV1 at Baseline and a minimum of 1 post-Baseline assessment before Week 8. Here, 'Number analyzed' signifies participants evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: days with interventions per study
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 116 | 116
days with interventions per study
  Hospitalization | 0.010 (0.0222) | 0.021 (0.0469)
  Use of Antibiotics | 0.220 (0.2284) | 0.245 (0.2380)

13. Other Pre Specified Outcome: Rate of Disruptions in Activities of Daily Living Because of Pulmonary Symptoms
Description: During treatment, any disruption in the activities of daily living, such as missed school or work, was documented if it was due to an exacerbation-like episode. Participants and caregivers recorded all disruptions in an electronic diary. The rate of disruptions was defined as the total days with disruptions to daily living divided by the total study duration.
Time Frame: Baseline up to EOT (Week 48)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: days with disruptions per study
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 116 | 116
days with disruptions per study | 0.037 (0.0550) | 0.047 (0.0755)

14. Other Pre Specified Outcome: Change From Baseline in Body Weight at Week 48
Description: Participants were weighed, and the weight was recorded at Baseline and then every 8 weeks during the treatment period. Baseline was the latest valid assessment prior to the treatment. A positive change from Baseline indicates that weight increased.
Time Frame: Baseline, EOT (Week 48)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 116 | 116
kg
  Baseline | 53.46 (13.941) | 56.01 (13.149)
  Change From Baseline: number analyzed (Participants) | 100 | 104
  Change From Baseline | 0.87 (3.342) | 0.83 (3.101)

15. Other Pre Specified Outcome: Change From Baseline in the Concentration of Interleukin-8 (IL-8) in Serum and Sputum at Week 48
Description: Expression of IL-8 was measured in serum and in sputum. Sputum was spontaneously produced and tested by using standardized procedures developed by the Cystic Fibrosis Foundation Therapeutics, Inc. Therapeutics Development Network (CFFT-TDN). Baseline was the latest valid assessment prior to the treatment. A negative change from Baseline indicates that the concentration of IL-8 decreased.
Time Frame: Baseline, EOT (Week 48)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: picograms/mL
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 116 | 116
picograms/mL
  Serum, Baseline: number analyzed (Participants) | 115 | 116
  Serum, Baseline | 39.537 (14.1697) | 55.845 (131.8505)
  Serum, Change From Baseline: number analyzed (Participants) | 96 | 103
  Serum, Change From Baseline | -2.334 (13.2141) | -16.197 (138.3108)
  Sputum, Baseline: number analyzed (Participants) | 94 | 95
  Sputum, Baseline | 267629.93 (259089.569) | 250170.95 (180581.976)
  Sputum, Change From Baseline: number analyzed (Participants) | 73 | 81
  Sputum, Change From Baseline | 28882.79 (199160.845) | 9957.24 (166348.660)

16. Other Pre Specified Outcome: Change From Baseline in the Concentration of Neutrophil Elastase in Sputum at Week 48
Description: Expression of neutrophil elastase was measured in sputum. Sputum was spontaneously produced and tested by using standardized procedures developed by the CFFT-TDN. Baseline was the latest valid assessment prior to the treatment. A positive change from Baseline indicates that the concentration of neutrophil elastase increased.
Time Frame: Baseline, EOT (Week 48)
Population: The ITT Population: all randomized participants with data for FEV1 at Baseline and a minimum of 1 post-Baseline assessment before Week 8. Here, 'Number analyzed' signifies participants evaluable for this outcome measure. Twenty-two participants each in the ataluren and placebo groups were not evaluable.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 94 | 94
ug/mL
  Baseline | 183.64 (221.901) | 227.35 (227.881)
  Change From Baseline: number analyzed (Participants) | 73 | 80
  Change From Baseline | 5.45 (232.824) | -8.67 (296.105)

17. Other Pre Specified Outcome: Change From Baseline in the Concentration of C-Reactive Protein (CRP) in Serum at Week 48
Description: Expression of CRP was measured in serum. Baseline was the latest valid assessment prior to the treatment. A positive change from Baseline indicates that CRP concentration increased.
Time Frame: Baseline, EOT (Week 48)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/liter (L)
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 116 | 116
mg/liter (L)
  Baseline: number analyzed (Participants) | 115 | 116
  Baseline | 6.899 (11.5869) | 7.037 (8.4411)
  Change From Baseline: number analyzed (Participants) | 96 | 103
  Change From Baseline | 2.420 (10.5162) | 2.031 (10.1202)

18. Other Pre Specified Outcome: Change From Baseline in the Total Lung Score as Assessed by Computed Tomography (CT) at Week 48
Description: Lungs were imaged by using non-contrast, spiral CT. The total lung score for each CT scan was established by the sum of 5 characteristics from the Brody scoring system, with scores ranging from 0 to 40.5, with lower scores indicating better lung function. The characteristics scored were bronchiectasis (score range 0 - 12), mucus plugging (score range 0- 6), peribronchial thickening (score range 0 - 9), parenchyma (score range 0 - 9), and hyperinflation (score range 0 - 4.5). Baseline was the latest valid assessment prior to the treatment. A positive change from Baseline indicates that lung function worsened.
Time Frame: Baseline, EOT (Week 48)
Population: The ITT Population: all randomized participants with data for FEV1 at Baseline and a minimum of 1 post-Baseline assessment before Week 8. Here, 'Number analyzed' signifies participants evaluable for this outcome measure. Eleven and 10 participants in the ataluren and placebo groups, respectively, were not evaluable.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 105 | 106
units on a scale
  Baseline | 9.531 (3.7526) | 9.619 (3.4244)
  Change From Baseline: number analyzed (Participants) | 99 | 104
  Change From Baseline | 0.282 (1.3441) | 0.560 (1.5602)

19. Other Pre Specified Outcome: Change From Baseline in Total Nasal Chloride Transport as Assessed by Transepithelial Potential Difference (TEPD) at Week 48
Description: TEPD was assessed in each nostril using standardized equipment, techniques, and solutions. Assessments were made on the nasal epithelium cells lining the inferior turbinate. Warmed solutions of Ringer's solution, amiloride, chloride-free gluconate, isoproterenol, and adenosine triphosphate (ATP) were perfused for ≥3-minute sequentially through a nasal catheter while a voltage tracing was recorded. Total chloride transport was computed for each nostril. The total chloride transport values were calculated by subtracting the voltages at the end of a perfusion from the voltage at the end of an earlier perfusion (isoproterenol - amiloride). The average of the values for each nostril was computed. If the assessment was available in only 1 nostril, this value was used as if it were the average of both nostrils. Baseline was the latest, valid assessment prior to the treatment. A positive change from Baseline indicates that nasal chloride transport increased.
Time Frame: Baseline, EOT (Week 48)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millivolts
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 116 | 116
millivolts
  Baseline | 1.578 (3.8786) | 1.950 (3.5462)
  Change From Baseline: number analyzed (Participants) | 100 | 104
  Change From Baseline | 0.312 (5.0574) | 0.139 (5.8139)

20. Other Pre Specified Outcome: Change From Baseline in Sweat Chloride Concentration at Week 48
Description: Sweat was collected, from each arm, by using pilocarpine iontophoresis. The chloride concentration in the sweat was quantified for each arm by using standard laboratory methods. Tests were also considered valid if the sweat collection time was ≤35 minutes; tests with longer collection times were also considered valid if extra time was needed to obtain sufficient volume (≥15uL) for analysis. For analysis purposes, the average of the values from each arm were computed. If the assessment was valid and/or available in only 1 arm, this value was used as if it were the average of both arms. The method used was consistent with the CFFT-TDN guidelines. Baseline was the latest, valid assessment prior to the treatment. A negative change from Baseline indicates that sweat chloride concentration decreased.
Time Frame: Baseline, EOT (Week 48)
Population: The ITT Population: all randomized participants with data for FEV1 at Baseline and a minimum of 1 post-Baseline assessment before Week 8. Here, 'Number analyzed' signifies participants evaluable for this outcome measure. Two and 5 participants in the ataluren and placebo groups, respectively, were not evaluable.
Measure: Mean (Standard Deviation); unit: millimoles/L
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 114 | 111
millimoles/L
  Baseline | 100.140 (14.2170) | 96.586 (15.9279)
  Change From Baseline: number analyzed (Participants) | 97 | 97
  Change From Baseline | -1.325 (8.9431) | -0.619 (10.2657)

ADVERSE EVENTS:
Time Frame: Baseline up to 4 Weeks Post-Treatment (Week 52) or Premature Discontinuation (PD)
Description: The As-Treated Population: all randomized participants who received at least 1 dose of study drug.
Arm/Group | Ataluren | Placebo
Serious Adverse Events (participants affected / at risk) | 46/120 | 50/118
Other Adverse Events (participants affected / at risk) | 118/120 | 115/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ataluren (N=120) | Placebo (N=118)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Drug withdrawal syndrome (General disorders) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia mycoplasmal (Infections and infestations) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Mycobacterium abscessus infection (Infections and infestations) | 0 (0) | 2 (2)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 3 (3) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 3 (3) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Cystic fibrosis long (Respiratory, thoracic and mediastinal disorders) | 34 (47) | 41 (66)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ataluren (N=120) | Placebo (N=118)
Abdominal pain (Gastrointestinal disorders) | 20 | 14
Vomiting (Gastrointestinal disorders) | 14 | 11
Diarrhoea (Gastrointestinal disorders) | 13 | 21
Abdominal pain upper (Gastrointestinal disorders) | 11 | 7
Nausea (Gastrointestinal disorders) | 11 | 13
Constipation (Gastrointestinal disorders) | 7 | 9
Pyrexia (General disorders) | 17 | 22
Fatigue (General disorders) | 11 | 11
Viral upper respiratory tract infection (Infections and infestations) | 21 | 32
Sinusitis (Infections and infestations) | 15 | 14
Rhinitis (Infections and infestations) | 12 | 13
Nasopharyngitis (Infections and infestations) | 10 | 8
Pharyngitis (Infections and infestations) | 7 | 4
Upper respiratory tract infection (Infections and infestations) | 5 | 12
Abnormal loss of weight (Metabolism and nutrition disorders) | 10 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 6
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 8 | 1
Headache (Nervous system disorders) | 20 | 14
Nephrolithiasis (Renal and urinary disorders) | 8 | 4
Dysuria (Renal and urinary disorders) | 7 | 1
Cystic fibrosis lung (Respiratory, thoracic and mediastinal disorders) | 85 | 82
Cough (Respiratory, thoracic and mediastinal disorders) | 28 | 35
Productive cough (Respiratory, thoracic and mediastinal disorders) | 12 | 11
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 9 | 16
Rales (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 14
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor can review results and/or communications prior to public release and can embargo communications regarding trial results for a period that is up to 180 days from the time submitted to the sponsor for review. The sponsor may consult with the PI to require changes to the communication or extend the embargo.